CLINICAL TRIAL: NCT05039073
Title: A Phase 2 Study of Brentuximab Vedotin Plus Nivolumab in Patients With Relapsed/Refractory Hodgkin Lymphoma Previously Treated With Brentuximab or Checkpoint Inhibitors
Brief Title: Brentuximab Vedotin and Nivolumab for the Treatment of Relapsed/Refractory Classic Hodgkin Lymphoma Previously Treated With Brentuximab Vedotin or Checkpoint Inhibitors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kristie Blum, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002348; NCI-2021-01655 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP5260-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-08-30; First posted 2021-09-09 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Classic Hodgkin Lymphoma; Refractory Classic Hodgkin Lymphoma
MeSH Terms: interventions — Brentuximab Vedotin; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (brentuximab vedotin, nivolumab) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 16 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response or partial response at any time after 4 cycles may discontinue study therapy to proceed to autologous or allogeneic stem cell transplant.
  Interventions: Drug: Brentuximab Vedotin; Procedure: Hematopoietic Cell Transplantation; Biological: Nivolumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Procedure: Hematopoietic Cell Transplantation — Undergo HSCT
  Other Names: HCT; Hematopoietic Stem Cell Infusion; Hematopoietic Stem Cell Transplantation; HSCT; Stem Cell Transplant; stem cell transplantation
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effect of brentuximab vedotin and nivolumab in treating patients with classic Hodgkin lymphoma that has come back (relapsed) or does not respond to treatment (refractory) that have been previously treated with brentuximab vedotin or checkpoint inhibitors. Brentuximab vedotin is a monoclonal antibody, brentuximab, linked to a toxic agent called vedotin. Brentuximab attaches to CD30 positive cancer cells in a targeted way and delivers vedotin to kill them. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving brentuximab vedotin and nivolumab in combination may be an effective treatment in patients with relapsed or refractory classic Hodgkin lymphoma previously treated with brentuximab vedotin or checkpoint inhibitors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR) with brentuximab vedotin (brentuximab)/nivolumab used in combination in patients in patients previously treated with brentuximab in combination with standard chemotherapy for Hodgkin lymphoma (HL).

II. To determine the ORR with brentuximab/nivolumab in combination in patients previously treated with checkpoint inhibitors alone or in combination with standard chemotherapy for HL.

SECONDARY OBJECTIVES:

I. To determine the complete response rate (CRR) and progression-free survival (PFS) with brentuximab/nivolumab in patients previously treated with brentuximab in combination with standard chemotherapy for HL.

II. To determine the CRR and PFS with brentuximab/nivolumab in patients previously treated with checkpoint inhibitors alone or in combination with standard chemotherapy for HL.

III. To evaluate safety of this regimen using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 (v 5.0).

IV. To determine the tolerability of this regimen using patient-reported outcomes including Patient Reported Outcomes (PRO)-CTCAE or pediatric PRO-CTCAE, neuropathy (Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity [FACT/GOG-NTX]), and fatigue quality of life (QOL) by strata.

V. To determine the number of patients who proceed to autologous or allogeneic hematopoietic stem cell transplantation (HSCT).

VI. To determine the number of patients who successfully undergo stem cell collection among those planning to proceed to autologous HSCT.

OUTLINE:

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes and nivolumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 16 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response or partial response at any time after 4 cycles may discontinue study therapy to proceed to autologous or allogeneic stem cell transplant.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed classical Hodgkin lymphoma
* Patients must be 12 years of age or older
* Patients must have received at least 1-2 prior multi-agent chemotherapy or immunotherapy regimens will be divided into two cohorts based on the following clinical scenarios:

  * Patients enrolled to cohort A must have received only ONE prior brentuximab-containing regimen with NO prior checkpoint inhibitors. Patients enrolled to cohort A must have received brentuximab as part of their first-line treatment regimen.
  * Patients enrolled to cohort B must have received only ONE prior immune checkpoint inhibitor- (i.e. nivolumab or pembrolizumab) containing regimen and NO prior brentuximab. Patients in cohort B may have received an immune checkpoint inhibitor during either their first- or second-line treatment regimen.
  * If radiation is used as part of the planned front-line treatment regimen (i.e., brentuximab vedotin-doxorubicin-vinblastine-dacarbazine [BV-AVD] + radiation therapy [RT] for bulky stage II disease), this will count as only 1 prior therapy. Additionally, radiation as consolidation after a second-line multi-agent chemotherapy regimen is permitted and will not be counted as a third regimen
* No prior autologous or allogeneic transplant
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 for patients > 18 years old, or Lansky performance status of >= 50 for patients ages 12-18 years
* Enrolling patients must have measurable disease defined as a tumor or nodal mass > 1.5 cm in at least one dimension
* Resolution of all prior toxicities, including peripheral neuropathy, to a =< grade 1
* Absolute neutrophil count (ANC) >= 750, unless disease related (within 28 days of cycle 1 day 1)
* Platelets >= 50,000, unless disease related (within 28 days of cycle 1 day 1)
* Creatinine =< upper limit of normal (ULN) (within 28 days of cycle 1 day 1)
* Aspartate aminotransferase/alanine aminotransferase (AST/ALT) =< 3 x ULN (within 28 days of cycle 1 day 1)
* Bilirubin =< 2 mg/dL (within 28 days of cycle 1 day 1)
* Patients with human immunodeficiency virus (HIV) infection are eligible. Patients with HIV infection must meet the following criteria: No evidence of co-infection with hepatitis B or C; CD4+ count >= 400/mm; no evidence of resistant strains of HIV; on anti-HIV therapy with an HIV viral load < 50 copies HIV ribonucleic acid (RNA)/mL. Patients with HIV must have ongoing follow-up with an infectious disease specialist and must have been evaluated within 90 days of cycle 1 day 1.
* Females of child-bearing potential (FCBP) must have a negative urine pregnancy test prior to starting therapy. If the test is positive, pregnancy must be ruled out
* FCBP and men treated or enrolled on this protocol must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry for the duration of study participation, and 6 months after completion of brentuximab and/or nivolumab administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

  * A female of childbearing potential (FCBP) is a post-menarcheal woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months
* Completion of all previous therapy (including surgery, radiotherapy, chemotherapy, immunotherapy, or investigational therapy) for the treatment of cancer >= 2 weeks before the start of study therapy
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions
* Evidence of a personally signed informed consent by patients >= 18 year old (YO) or parent or legally authorized representative (LAR) for patients 12-17 YO indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation. Patients 12-17 will also be required to give assent to the process per institutional guidelines

Exclusion Criteria:

* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for >= 2 years or which will not limit survival to < 2 years
* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events to =< grade 1
* Active autoimmune disease or history of autoimmune disease such as hepatitis, hypophysitis, nephritis, interstitial lung disease, and colitis
* Active central nervous system (CNS) involvement with lymphoma
* Patients with hepatitis B (positive hepatitis B virus surface antigen [HBsAg] or hepatitis B virus core antibody [HBcAb]) and those with positive hepatitis C virus (HCV) antibodies are not permitted to enroll
* No active infection, or other active illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 16 cycles (each cycle is 21 days)
  Will be calculated and a 95% confidence interval will be estimated using the Clopper-Pearson method. Assessed per Lugano 2014 Criteria at any time point while on study therapy. Will be analyzed independently for each cohort (A and B).

SECONDARY OUTCOMES:
Complete response rate (CRR) | Up to 16 cycles (each cycle is 21 days)
  Will be calculated and a 95% confidence interval will be estimated using the Clopper-Pearson method. Will be determined per Lugano 2014 criteria at any disease assessment time point while the patient is receiving study therapy.
Progression-free survival (PFS) | From time of study enrollment until first documentation of progressive disease or death from any cause, assessed up to 5 years
  Will be described using the Kaplan-Meier methodology. 95% confidence intervals for 1-year and 2-year PFS will be calculated, with standard errors estimated using the Greenwood formula. Patients alive without disease progression will be censored at last follow-up date.
Overall survival (OS) | From time of study enrollment until death from any cause, assessed up to 5 years
  Will be described using the Kaplan-Meier methodology. 95% confidence intervals for 1-year and 2-year OS will be calculated, with standard errors estimated using the Greenwood formula. Patients who have not died will be censored at last follow-up date.
Incidence of adverse events | Up to 5 years
  According to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0).
Incidence of symptomatic toxicity | Up to 5 years
  Evaluated by Patient Reported Outcomes (PRO)-CTCAE or Pediatric PRO-CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Blum, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No